CLINICAL TRIAL: NCT03018015
Title: Characterisation of Relative Bioavailability of a Newly Developed Ibuprofen Oral Powder Formulation in Comparison With Two Marketed Reference Products in a Single Dose, 3-period-crossover Design Under Fasting Conditions; Controlled, Open-label, Randomised Study With Bioequivalence Assessment
Brief Title: Ibuprofen Bioavailability Trial With Oral Single Dose Administration.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SocraTec R&D GmbH (Other)
Collaborators: SocraMetrics GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 1325ib16ct
Record Dates: First submitted 2017-01-10; First posted 2017-01-11 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Bioequivalence
Keywords: Bioequivalence; Healthy; Bioavailability; Ibuprofen
MeSH Terms: interventions — Ibuprofen; Powders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ibuprofen 400 mg oral powder (Experimental): oral fasted administration of 1 sachet of Ibuprofen 400 mg oral powder (Hermes Arzneimittel GmbH, Germany), containing 400 mg ibuprofen
  Interventions: Drug: Ibuprofen 400 mg oral powder
- Brufen 400 mg film-coated tablets (Active Comparator): oral fasted administration of Brufen 400 mg film-coated tablets (Abbott Scandinavia AB, Sweden), containing 400 mg ibuprofen
  Interventions: Drug: Ibuprofen 400 mg film-coated tablet
- Spalt forte 400 mg Weichkapseln (Active Comparator): oral fasted administration of Spalt forte 400 mg Weichkapseln (Pfizer Consumer Healthcare GmbH, Germany), containing 400 mg ibuprofen
  Interventions: Drug: Ibuprofen 400 mg soft capsule

INTERVENTIONS:
Drug: Ibuprofen 400 mg oral powder
  Arms: Ibuprofen 400 mg oral powder
Drug: Ibuprofen 400 mg film-coated tablet
  Arms: Brufen 400 mg film-coated tablets
Drug: Ibuprofen 400 mg soft capsule
  Arms: Spalt forte 400 mg Weichkapseln

SUMMARY:
The present study will be conducted in order to assess bioequivalence of the Test product (Ibuprofen 400 mg oral powder) and the Reference product 1 (Brufen 400 mg film-coated tablet), an approved market product in the European Union. Testing for bioequivalence will be performed considering AUC0-tlast and Cmax obtained after oral single dose fasted administration of ibuprofen.

In addition to the conventional immediate release tablet used as Reference 1, a soft capsule formulation will be applied as Reference 2 (Spalt Forte 400 mg Weichkapseln), as an example for a product with a very fast absorption rate.

All 3 immediate release preparations contain 400 mg ibuprofen.

DETAILED DESCRIPTION:
The clinical trial will be performed in a single centre, open-label, randomised (order of treatments), balanced, 3-period, 6-sequence, single dose change-over design with administration under fasting conditions separated by a washout period of at least 2 treatment-free days.

Blood sample collection will be performed over 16 h after administration. This time is considered adequate to characterise plasma concentration vs. time profiles long enough for reliable estimation of the extent of absorption, i.e. the AUC derived from measurements is expected to cover at least 80 % of the AUC extrapolated to infinity.

ELIGIBILITY:
Inclusion Criteria:

1. sex: male/female
2. ethnic origin: Caucasian
3. age: 18 years or older
4. body-mass index (BMI): ≥ 18.5 kg/m² and ≤ 30.0 kg/m², body weight > 40 kg
5. good state of health
6. non-smoker or ex-smoker for at least 3 months
7. written informed consent, after having been informed about benefits and potential risks of the clinical trial, as well as details of the insurance taken out to cover the subjects participating in the clinical trial

Exclusion Criteria:

1. existing cardiac and/or haematological diseases or pathological findings, which might interfere with the safety or tolerability of the active ingredient
2. existing hepatic and/or renal diseases or pathological findings, which might interfere with the safety or tolerability, and/or pharmacokinetics of the active ingredient
3. existing gastrointestinal diseases or pathological findings, which might interfere with the safety, tolerability, absorption and/or pharmacokinetics of the active ingredient
4. history of gastrointestinal bleeding or perforation, related to previous NSAID therapy
5. existing, or history of, recurrent gastrointestinal ulcer/ bleeding
6. conditions involving an increased tendency to bleeding
7. active or known inflammatory bowel diseases (e.g. colitis ulcerosa, Crohn´s disease)
8. history of relevant CNS and/or psychiatric disorders and/or currently treated CNS and/or psychiatric disorders
9. known allergic reactions to the active ingredients used or to constituents of the pharmaceutical preparations
10. history of hypersensitivity reactions (e.g. bronchial spasm, asthma, rhinitis, urticaria, or angioedema) after intake of acetylsalicylic acid or other NSAIDs
11. subjects with severe allergies or multiple drug allergies unless it is judged as not relevant for the clinical trial by the investigator
12. existing, or history of, bronchial asthma, chronic rhinitis or allergic diseases unless it is judged as not relevant for the clinical trial by the investigator
13. subjects with hereditary problems of galactose intolerance, lactase deficiency or glucose-galactose malabsorption
14. systolic blood pressure < 90 or > 145 mmHg
15. diastolic blood pressure < 60 or >90 mmHg
16. heart rate < 50 bpm or > 90 bpm
17. laboratory values out of normal range unless the deviation from normal is judged as not relevant for the clinical trial by the investigator except parameters ASAT, ALAT, bilirubin and creatinine (see exclusion criterion No. 18)
18. laboratory values: ASAT > 20 % ULN, ALAT > 10 % ULN, bilirubin > 20 % ULN and creatinine > 9 μmol/l ULN
19. positive anti-HIV-test (if positive to be verified by western blot), HBs-AG-test (if positive to be verified by test for HBc-IgM) or anti-HCVtest
20. acute or chronic diseases which may interfere with the pharmacokinetics of the IMP
21. history of or current drug or alcohol dependence
22. positive alcohol or drug test at screening examination
23. regular intake of alcoholic food or beverages of ≥ 40 g pure ethanol for male or ≥ 20 g pure ethanol for female per day
24. subjects who are on a diet which could affect the pharmacokinetics of the active ingredient
25. regular intake of caffeine containing food or beverages of ≥ 500 mg caffeine per day
26. blood donation or other blood loss of more than 400 ml within the last 2 months prior to individual enrolment of the subject
27. administration of any investigational medicinal product during the last 2 months prior to individual enrolment of the subject
28. regular treatment with any systemically available medication (except hormonal contraceptives)
29. subjects, who report a frequent occurrence of migraine attacks
30. positive pregnancy test at screening examination
31. pregnant or lactating women
32. female subjects who do not agree to apply highly effective contraceptive methods
33. subjects suspected or known not to follow instructions
34. subjects who are unable to understand the written and verbal instructions, in particular regarding the risks and inconveniences they will be exposed to during their participation in the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-09; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC0-tlast) for ibuprofen | 16 hours interval
Peak Plasma Concentration (Cmax) for ibuprofen | 16 hours interval

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events | from first dose until discharge of the subject (approx. 2 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Cornelius Koch, MD, Principal Investigator — SocraTec R&D GmbH, Clinical Pharmacology Unit
Locations (1):
- SocraTec R&D GmbH Clinical Pharmacology Unit, Erfurt, Thuringia, Germany